CLINICAL TRIAL: NCT06863883
Title: Measuring Outcomes in Aortic STenosis Patients Undergoing AVR - Evaluation of Prognosis Regarding Short- and Long-term Results (MASTER)
Brief Title: Aortic Stenosis - Prognosis, Risk and Outcomes
Acronym: MASTER
Status: Not yet recruiting | Type: Observational
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Other Study IDs: EPM Dnr 2024-06746-01
Record Dates: First submitted 2025-01-13; First posted 2025-03-07 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-02

CONDITIONS: Aortic Stenosis Disease
Keywords: TAVI; Cardiac remodelling; Aortic stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples for metabolomics , proteomics and circulating miRNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- TAVI patients: 300 patients undergoing TAVI at Sahlgrenska University Hospital

SUMMARY:
The investigators will prospectively enroll 300 patients undergoing TAVI at Sahlgrenska University Hospital, which is the second largest TAVI hospital in Sweden. Eligible patients should have a clinical indication for aortic valve replacement with TAVI and have preprocedural clinical investigations with echocardiography (UCG) and CCT and provide written informed consent. UCG, electrocardiogram (ECG) and blood samples will be taken in addition to clinical status, NYHA-class and collection of outcome events the day before the procedure, 1±2 hours, 24 ±6hours and daily after the procedure until discharged from Sahlgrenska. Further follow-up will be scheduled day 14, 30, 180, 365 and yearly. Cardiac MRI will be performed before, at 14 days and at 180 days after TAVI. Brain MRI will be performed before and 24± hours after TAVI. Cardiac CT will be performed at 180 days after TAVI.

DETAILED DESCRIPTION:
* Study procedures UCG, cardiac CT and ECG before the TAVI procedure are done as standard of care. Study-related imaging procedures are non-invasive methods that carry no risk of serious adverse events for the study subject.
* Ultrasound cardiogram (UCG) UCG is a non-invasive imaging procedure that uses ultrasound to image the heart in real- time. UCG carries no risk of causing serious adverse events for the study participants.
* Quality of life Quality of life will be assessed using EQ-5D-5L at baseline and at 14 days, 30 days, 180 days and yearly after the procedure.
* ECG ECG has been the cornerstone of cardiovascular medicine for decades and is part of routine clinical practice for all patients undergoing TAVI at cardiology departments across the world. It is a non-invasive test that carries no risk of serious adverse events.
* MRI Cardiac Magnetic Resonance imaging (CMR) will be used to assess the degree of cardiac remodeling and hemodynamic and blood flow parameters, e.g. turbulence, as a sub-study within in the larger study. Brain Magnetic Resonance imaging (brain MRI) will be used to assess micro-embolism and ischemic stroke related to the TAVI procedure.

CMR and Brain MRI poses no increased risk of causing serious adverse events for patients participating in the study. However, patients with clear contraindication will not be included to the study. (e.g. patients with MRI non-compatible metal device present in body, claustrophobia or for other reasons set at the local clinic). Patients with kidney failure (estimated glomerular filtration rate <30 ml/kg/min,) will not be given MRI contrast medium.

MRI is planned before the TAVI procedure (baseline), 24 hours (Brain MRI) and at 180 days (CMR) after TAVI.

* Cardiac CT Cardiac CT before TAVI is part of routine clinical care and used for procedural planning. An additional cardiac CT will be performed as a sub-study at 180 days after the TAVI procedure. The procedure will be used to assess the placement of the TAVI-valve in the native aortic annulus, e.g. the depth of the valve, the alignment of the commissures of the prothesis in relation the native commissures and the coronary ostia and be used to simulate the possibilities to perform a redo-TAVI if the need should arise. Patients with kidney failure (estimated glomerular filtration rate <30 ml/kg/min,) will not be given CT contrast medium.
* Storing of blood samples for future analysis Plan to save blood samples (for subjects that have consented to this part) for the purpose of future analysis for metabolomics, proteomics and circulating miRNA. The amount of blood for biobank storage will be 21 ml collected at four time points per study participant, i.e. max 84 ml per patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient with clinical indication for aortic valve replacement and scheduled for TAVI
* Patient willing and able to provide signed informed consent

Exclusion Criteria:

* Inability to provide informed consent Additional exclusion criteria for MRI
* Estimated glomerular filtration rate <30 ml/kg/min (MRI without contrast can be performed )
* Claustrophobia or inability to tolerate confined spaces.
* Non-compatible metal device present in body
* Any other contra-indications for MRI as per local guidelines Additional exclusion criteria for the CT substudy
* Estimated glomerular filtration rate <30 ml/kg/min (CT without contrast can be performed)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: We will prospectively enroll 300 patients undergoing TAVI at Sahlgrenska University Hospital
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2030-12 (Estimated); Study Completion 2031-06 (Estimated)

PRIMARY OUTCOMES:
Cardiac damage | Baseline and 180 days
  To study change in stage of cardiac damage (stage 0-4) by echocardiography.

SECONDARY OUTCOMES:
Change in echocardiography parameters | Baseline and at 14, 30 and 180 days
  To study E/é ratio in echocardiography derived parameters indicating cardiac damage (delta%)
Change in echocardiography parameters | Baseline and at 14, 30 and 180 days
  To study Left ventricular mass change on echocardiography (delta gram)
Left Atrial -strain | Baseline and at 14, 30 and 180 days
  To study change in LA-strain derived by echocardiography (delta %)
Change in echocardiography parameters | Baseline and at 14, 30 and 180 days
  To study the influence of effectiv orfice area (cm2)of the aortic valve on cardiac damage (stage 0-4)
Cardiac Magnetic Resonance (CMR) | Baseline and at 14 and 180 days
  Change in CMR derived parameters Left ventricular mass (delta gram)

CONTACTS AND LOCATIONS:
Locations (1):
- Departement of Cardiology, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No